CLINICAL TRIAL: NCT00951938
Title: A Radiographic and Clinical Study Evaluating a Novel Allogeneic, Cancellous, Bone Matrix Containing Viable Stem Cells (Trinity Evolution™ Viable Cryopreserved Cellular Bone Matrix) in Patients Undergoing Anterior Cervical Discectomy and Fusion
Brief Title: Trinity Evolution in Anterior Cervical Disectomy and Fusion (ACDF)
Status: Completed | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-01005A
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Degenerative Disc Disease
Keywords: Trinity Evolution; Anterior Cervical Discectomy and Fusion; Allograft
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to utilize Trinity Evolution in conjunction with an interbody spacer and supplemental anterior fixation of the surgeon's choice and to follow the patients to measure the clinical outcomes and rate of fusion. The hypothesis of the study is that Trinity Evolution combined with an interbody spacer and supplemental anterior fixation will result in fusion rates and clinical outcomes similar to those with other routinely used autograft and allograft materials including: fusion, improvement in pain and function, maintenance of upper extremity neurological function, and absence of serious adverse events related to the use of the Trinity Evolution product.

DETAILED DESCRIPTION:
When conservative care fails to alleviate the pain and neurological deficits caused by degenerative disc disease in a cervical spine, the most common recourse is surgical decompression of the affected nerves and/or spinal cord. Decompression is often accomplished via an anterior approach whereby essentially the entire disc as well as any bony osteophytes and ligaments that are compressing the spinal cord and/or nerves are removed. While usually successful at decompressing affected neural structures, the decompression often results in collapse of the disc space, instability and recurrent symptomatology.

Most anterior cervical decompressions therefore are followed by insertion of a structural interbody spacer such as a bone graft from the patient's iliac crest (autograft) or a bone graft from a cadaver (allograft). The "gold standard" for aiding healing in spinal fusion surgeries is the harvesting of autograft from the patient's iliac crest and placing it in and around the segments of the spine that are intended to be fused. Autograft is considered the "gold standard" because it contains the essential elements required for successful bone grafting: osteogenesis, osteoconduction, and osteoinduction.

However, the morbidity of harvesting autograft has been well documented and includes chronic donor-site pain, infection, neurologic injury, blood loss, deformity, bowel injury, hernia, and prolonged surgical and hospitalization time. There are now a number of products on the market to minimize or replace the use of autograft. However, few of these products contain all three essential bone-forming elements (osteogenesis, osteoconduction, and osteoinduction) in a single, stand alone product.

Trinity Evolution is a novel, allogeneic cancellous bone matrix containing viable osteoprogenitor cells, mesenchymal stem cells and demineralized cortical bone (DCB) component to provide the required osteoconduction, osteogenesis, and osteoinduction necessary for successful bone grafting. Preclinical studies with Trinity Evolution have demonstrated in-vitro and in-vivo safety and effectiveness. Trinity Evolution is considered an allograft and as such is a "minimally manipulated" tissue and is labeled for bone repair for spinal, orthopedic and podiatric indications where autograft is used. The dosage will be dependent upon the specific requirements of the case.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cervical degenerative disc disease at up to four levels between C3 and T1
* Neck and/or arm pain and/or a functional neurological deficit, and/or cervical myelopathy with neural compression confirmed by plain x-rays and MRI, Myelogram or CT. Scheduled for an ACDF with a spacer and anterior supplemental fixation of the surgeon's choice.
* Greater than 18 years of age
* Unresponsive to conservative care over a period of at least 6 weeks or has progressive neurological signs and/or symptoms of neurological compromise that mandate urgent surgical intervention.
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent.

Exclusion Criteria:

* More than 4 levels (C3 - T1) requiring surgical treatment
* Active local or systemic infection
* Currently pregnant or considering becoming pregnant during the follow-up period
* Active malignancy or having been on chemotherapy of any kind for a malignancy in the past 1 year.
* Axial neck pain as the primary diagnosis, without evidence of neural compression
* Use of any other bone graft or bone graft substitute in addition to or in place of Trinity Evolution in and around the interbody spacer
* Use of adjunctive post-operative stimulation
* Prior interbody surgery at the same level
* Has a known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will be conducted by patient's neurosurgeon or orthopedic surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fusion Rates for Trinity Evolution | Operative to 12 months Follow-up

SECONDARY OUTCOMES:
NDI relative improvement, VAS improvement, Maintenance or improvement of neurological function | Pre-operative to 12 months follow-up
Complication Rates for Trinity Evolution | Operative to 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J Linovitz, MD, Study Director — Orthofix Spinal Implants
Locations (13):
- United States (13):
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Shasta Orthopaedics Spine Center, Redding, California
  - Denver-Vail Orthopedics, P.C., Parker, Colorado
  - Central Connecticut Neurosurgery and Spine, New Britain, Connecticut
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Michigan, A. Alfred Taubman Health Care Center, Ann Arbor, Michigan
  - Western Regional Center for Spine and Brain Surgery, Las Vegas, Nevada
  - Carolina NeuroSurgery & Spine, Charlotte, North Carolina
  - Triangle Neurosurgery, Raleigh, North Carolina
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Greater Houston Neurosurgery Center, The Woodlands, Texas
  - The Virginia Spine Institute, Reston, Virginia
  - Tuckahoe Orthopaedic Associates, Richmond, Virginia

REFERENCES:
- [Derived] Peppers TA, Bullard DE, Vanichkachorn JS, Stanley SK, Arnold PM, Waldorff EI, Hahn R, Atkinson BL, Ryaby JT, Linovitz RJ. Prospective clinical and radiographic evaluation of an allogeneic bone matrix containing stem cells (Trinity Evolution(R) Viable Cellular Bone Matrix) in patients undergoing two-level anterior cervical discectomy and fusion. J Orthop Surg Res. 2017 Apr 26;12(1):67. doi: 10.1186/s13018-017-0564-5. PMID 28446192